CLINICAL TRIAL: NCT03068520
Title: Imaging After Stereotactic Radiosurgery for Brain Metastases or Primary Tumor Can Hybrid PET-MRI Differentiate Between Radiation Effects and Disease ?
Brief Title: Can Hybrid PET-MRI Differentiate Between Radiation Effects and Disease Progression?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assuta Medical Center (Other)
Collaborators: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Michal Guindy, Medical Director of Imaging Services, Assuta Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 022-16-ASMC
Record Dates: First submitted 2017-02-20; First posted 2017-03-03 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Brain Tumor
Keywords: PET; MRI; BRAIN METASTASIS; BRAIN PRIMARY TUMOR; RESPONSE TO TREATMENT
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: to use the combined data obtained by PET-MRI scanning regarding amino acid metabolic profile, functional and morphological details in order to:
  1. Distinguish between progressive tumor and treatment related effects
  2. To identify pseudoresponse to antiangiogenic therapy from tumor progression
  3. To optimize the study protocol of PET-MRI for future routine clinical application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRIMARY BRAIN TUMOR (PBT) (Other): patients with PBT (Glioblastoma, Anaplastic Astrocytoma, Anaplastic Oligodendroglioma, Anaplastic Oligoastrocytoma), before treatment with radiation and chemotherapy.will be followed with PET MRI
  Interventions: Diagnostic Test: PET MR
- METASTATIC BT TREATED BY SRS (Other): patients with lung or breast metastasis to brain treated by SRS in which at least one lesion showed deterioration by MR performed after treatment.
  will be followed with PET MRI
  Interventions: Diagnostic Test: PET MR
- METASTATIC BT NOT TREATED BY SRS (Other): patients with lung or breast metastasis to brain where the SRS treatment was postponed for clinical reasons (getting mutation information for targeted treatment) the lesion size measures 5-40 mm.
  will be followed with PET MRI
  Interventions: Diagnostic Test: PET MR

INTERVENTIONS:
Diagnostic Test: PET MR — PET MR with 18 Fluorodopa ([18F]-DOPA) will be performed on patient at set intervals

SUMMARY:
PET-MRI scanning regarding amino acid metabolic profile, functional and morphological details will be performed on set intervals to patients with brain tumor & brain metastases in order to try to optimize the study protocol, distinguish between pseudo-response to anti-angiogenic therapy and tumor progression, and most importantly try to distinguish between progressive tumor and treatment related effects.3 cohort of patients will be included in the study.

DETAILED DESCRIPTION:
The multimodality approach for management of primary and secondary brain tumors includes surgery, radiotherapy and chemotherapy. Determination of an objective response to treatment relies on imaging findings (e.g. CT, MRI, PET).During the course of the disease patients with brain tumors often develop new or worsening contrast-enhancing lesions on routine follow-up imaging.These lesions may reflect tumor recurrence, treatment effect, or a combination of both. Discerning between tumor recurrence and treatment effect is clinically significant issue and a major challenge in neuro-oncology. Treatment-related effects exist within a spectrum, with "pseudoprogression" reflecting subacute and often transient injury, and "radiation necrosis" reflecting later and more permanent damage.The difficulty in differentiating tumor progression from treatment-related effects has serious implications for individual patient treatment decisions and prognosis as well as for clinical trial design and interpretation of results.

A contemporary hybrid scanner technology is capable of acquiring both metabolic information from PET and morphological and functional details from MRI. This new integrated technique opens new horizons for clinical and research evaluation of brain tumors and the associated treatment effects.

The aim of the current study is to use the combined data obtained by PET-MRI scanning regarding amino acid metabolic profile, functional and morphological details in order to:

1. Distinguish between progressive tumor and treatment related effects
2. To identify pseudo-response to antiangiogenic therapy from tumor progression
3. To optimize the study protocol of PET-MRI for future routine clinical application.

The study will include three cohorts of patients with brain tumors:

1. Primary brain tumors:

   A cohort of 60 adult patients (age: 18-70) with newly diagnosed high grade gliomas (Glioblastoma, Anaplastic Astrocytoma, Anaplastic Oligodendroglioma, Anaplastic Oligoastrocytoma) scheduled for a combined treatment with chemotherapy and radiotherapy. Patients will be eligible for the study immediately after receiving the pathological diagnosis and prior to any further treatment. These patients will undergo the PET-MRI scanning at 4 time points as follows:
   * 1st scan: after surgery or biopsy and before any further treatment
   * 2nd scan: will be performed up to 4 weeks after completing the combined radiotherapy and chemotherapy regimen.
   * 3rd and 4th scans: will follow with interval of 3 months between studies.
   * Additional scans will be performed by the decision of the investigators or when the patient is scheduled for antiangiogenic therapy
2. Brain metastases treated with stereotactic radiosurgery (SRS):

   A cohort of 60 adult patients (age: 18-75) who are being followed after SRS treatment for brain metastases secondary to breast or lung cancer whose recent imaging showed signs of progression in at list one of the previously treated lesion. Progression will be determined by Response Assessment in Neuro-Oncology Criteria (RANO criteria) for brain metastases. Number of target lesions should not exceed 4 with size of lesions ranging between 5-40 mm. These patients will undergo the PET-MRI scanning at three time points as follows:
   * 1st scan: Following determination of progression of SRS treated lesion based on standard surveillance MRI
   * 2nd and 3rd scans: will be performed every 2 months after the first scan
   * Additional scans will be performed by the decision of the investigators
3. Brain metastases not treated with SRS/radiotherapy

A cohort of 20 adult patients (age: 18-75) with a diagnosis of brain metastases secondary to human epidermal growth factor receptor 2 (HER2) positive breast cancer or anaplastic lymphoma kinase (ALK) or Epidermal Growth Factor Receptor (EGFR) gene mutant lung cancer who might be candidate for SRS treatment and in whom targeted therapy is selected instead. The size of the lesions should range between 5-40 mm. These patients will undergo the PET-MRI scanning at three time points as follows:

* 1st scan: after the first documentation of brain metastases on standard MRI
* 2nd and 3rd scans: will be performed every 2 months after the first scan
* In case of progression and SRS treatment follow-up scanning will be performed every 2 months
* Additional scans will be performed by the decision of the investigators

ELIGIBILITY:
Inclusion Criteria:

* Subject with glial brain tumors,
* Subjects with metastatic brain tumors that were treated with stereotactic radiation (SRS), * Subjects with metastatic brain tumors which were not treated

Exclusion Criteria:

* glial tumor with no histological diagnosis
* non breast of lung metastasis
* non compliance
* unable to lay still during the scanning
* mri non
* renal failure/gadolinium sensitivity
* less than 5 mm metastatic tumors
* bleeding brain tumors
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Distinguish between progressive tumor and treatment related effects | 1st scan: after surgery or biopsy and before any further treatment - 2nd scan: up to 4 weeks after completing the combined radiotherapy and chemotherapy regimen. - 3rd and 4th scans - 3 month interval apart
  finding PET-MRI difference between progression and treatment effect correlating with clinical out come

CONTACTS AND LOCATIONS:
Overall Officials: Michal Guindy, MD, Principal Investigator — Assuta Medical Center
Locations (1):
- Assuta Medical Centers, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horky LL, Treves ST. PET and SPECT in brain tumors and epilepsy. Neurosurg Clin N Am. 2011 Apr;22(2):169-84, viii. doi: 10.1016/j.nec.2010.12.003. PMID 21435569
- [Background] Chen W, Silverman DH, Delaloye S, Czernin J, Kamdar N, Pope W, Satyamurthy N, Schiepers C, Cloughesy T. 18F-FDOPA PET imaging of brain tumors: comparison study with 18F-FDG PET and evaluation of diagnostic accuracy. J Nucl Med. 2006 Jun;47(6):904-11. PMID 16741298
- [Background] Momose T, Nariai T, Kawabe T, Inaji M, Tanaka Y, Watanabe S, Maehara T, Oda K, Ishii K, Ishiwata K, Yamamoto M. Clinical benefit of 11C methionine PET imaging as a planning modality for radiosurgery of previously irradiated recurrent brain metastases. Clin Nucl Med. 2014 Nov;39(11):939-43. doi: 10.1097/RLU.0000000000000561. PMID 25140562
- [Background] Nanni C, Fanti S, Rubello D. 18F-DOPA PET and PET/CT. J Nucl Med. 2007 Oct;48(10):1577-9. doi: 10.2967/jnumed.107.041947. No abstract available. PMID 17909255
- [Background] Verma N, Cowperthwaite MC, Burnett MG, Markey MK. Differentiating tumor recurrence from treatment necrosis: a review of neuro-oncologic imaging strategies. Neuro Oncol. 2013 May;15(5):515-34. doi: 10.1093/neuonc/nos307. Epub 2013 Jan 16. PMID 23325863
- [Background] Tudisca C, Nasoodi A, Fraioli F. PET-MRI: clinical application of the new hybrid technology. Nucl Med Commun. 2015 Jul;36(7):666-78. doi: 10.1097/MNM.0000000000000312. PMID 25830717
- [Background] Kondziolka D, Patel A, Lunsford LD, Kassam A, Flickinger JC. Stereotactic radiosurgery plus whole brain radiotherapy versus radiotherapy alone for patients with multiple brain metastases. Int J Radiat Oncol Biol Phys. 1999 Sep 1;45(2):427-34. doi: 10.1016/s0360-3016(99)00198-4. PMID 10487566
- [Background] Aoyama H, Shirato H, Tago M, Nakagawa K, Toyoda T, Hatano K, Kenjyo M, Oya N, Hirota S, Shioura H, Kunieda E, Inomata T, Hayakawa K, Katoh N, Kobashi G. Stereotactic radiosurgery plus whole-brain radiation therapy vs stereotactic radiosurgery alone for treatment of brain metastases: a randomized controlled trial. JAMA. 2006 Jun 7;295(21):2483-91. doi: 10.1001/jama.295.21.2483. PMID 16757720
- [Background] Andrews DW, Scott CB, Sperduto PW, Flanders AE, Gaspar LE, Schell MC, Werner-Wasik M, Demas W, Ryu J, Bahary JP, Souhami L, Rotman M, Mehta MP, Curran WJ Jr. Whole brain radiation therapy with or without stereotactic radiosurgery boost for patients with one to three brain metastases: phase III results of the RTOG 9508 randomised trial. Lancet. 2004 May 22;363(9422):1665-72. doi: 10.1016/S0140-6736(04)16250-8. PMID 15158627
- [Background] Chang EL, Wefel JS, Hess KR, Allen PK, Lang FF, Kornguth DG, Arbuckle RB, Swint JM, Shiu AS, Maor MH, Meyers CA. Neurocognition in patients with brain metastases treated with radiosurgery or radiosurgery plus whole-brain irradiation: a randomised controlled trial. Lancet Oncol. 2009 Nov;10(11):1037-44. doi: 10.1016/S1470-2045(09)70263-3. Epub 2009 Oct 2. PMID 19801201
- [Background] Kocher M, Soffietti R, Abacioglu U, Villa S, Fauchon F, Baumert BG, Fariselli L, Tzuk-Shina T, Kortmann RD, Carrie C, Ben Hassel M, Kouri M, Valeinis E, van den Berge D, Collette S, Collette L, Mueller RP. Adjuvant whole-brain radiotherapy versus observation after radiosurgery or surgical resection of one to three cerebral metastases: results of the EORTC 22952-26001 study. J Clin Oncol. 2011 Jan 10;29(2):134-41. doi: 10.1200/JCO.2010.30.1655. Epub 2010 Nov 1. PMID 21041710
- [Background] Sahgal A. Point/Counterpoint: Stereotactic radiosurgery without whole-brain radiation for patients with a limited number of brain metastases: the current standard of care? Neuro Oncol. 2015 Jul;17(7):916-8. doi: 10.1093/neuonc/nov087. No abstract available. PMID 26092877
- [Background] Patel TR, McHugh BJ, Bi WL, Minja FJ, Knisely JP, Chiang VL. A comprehensive review of MR imaging changes following radiosurgery to 500 brain metastases. AJNR Am J Neuroradiol. 2011 Nov-Dec;32(10):1885-92. doi: 10.3174/ajnr.A2668. Epub 2011 Sep 15. PMID 21920854
- [Background] Ross DA, Sandler HM, Balter JM, Hayman JA, Archer PG, Auer DL. Imaging changes after stereotactic radiosurgery of primary and secondary malignant brain tumors. J Neurooncol. 2002 Jan;56(2):175-81. doi: 10.1023/a:1014571900854. PMID 11995819
- [Background] Walker AJ, Ruzevick J, Malayeri AA, Rigamonti D, Lim M, Redmond KJ, Kleinberg L. Postradiation imaging changes in the CNS: how can we differentiate between treatment effect and disease progression? Future Oncol. 2014 May;10(7):1277-97. doi: 10.2217/fon.13.271. PMID 24947265
- [Background] Kohutek ZA, Yamada Y, Chan TA, Brennan CW, Tabar V, Gutin PH, Yang TJ, Rosenblum MK, Ballangrud A, Young RJ, Zhang Z, Beal K. Long-term risk of radionecrosis and imaging changes after stereotactic radiosurgery for brain metastases. J Neurooncol. 2015 Oct;125(1):149-56. doi: 10.1007/s11060-015-1881-3. Epub 2015 Aug 26. PMID 26307446
- [Background] Sneed PK, Mendez J, Vemer-van den Hoek JG, Seymour ZA, Ma L, Molinaro AM, Fogh SE, Nakamura JL, McDermott MW. Adverse radiation effect after stereotactic radiosurgery for brain metastases: incidence, time course, and risk factors. J Neurosurg. 2015 Aug;123(2):373-86. doi: 10.3171/2014.10.JNS141610. Epub 2015 May 15. PMID 25978710
- [Background] Lin NU, Lee EQ, Aoyama H, Barani IJ, Barboriak DP, Baumert BG, Bendszus M, Brown PD, Camidge DR, Chang SM, Dancey J, de Vries EG, Gaspar LE, Harris GJ, Hodi FS, Kalkanis SN, Linskey ME, Macdonald DR, Margolin K, Mehta MP, Schiff D, Soffietti R, Suh JH, van den Bent MJ, Vogelbaum MA, Wen PY; Response Assessment in Neuro-Oncology (RANO) group. Response assessment criteria for brain metastases: proposal from the RANO group. Lancet Oncol. 2015 Jun;16(6):e270-8. doi: 10.1016/S1470-2045(15)70057-4. Epub 2015 May 27. PMID 26065612
- [Background] O'Brien BJ, Colen RR. Post-treatment imaging changes in primary brain tumors. Curr Oncol Rep. 2014;16(8):397. doi: 10.1007/s11912-014-0397-x. PMID 24997979
- [Background] Linhares P, Carvalho B, Figueiredo R, Reis RM, Vaz R. Early Pseudoprogression following Chemoradiotherapy in Glioblastoma Patients: The Value of RANO Evaluation. J Oncol. 2013;2013:690585. doi: 10.1155/2013/690585. Epub 2013 Aug 13. PMID 24000284
- [Background] Brandes AA, Franceschi E, Tosoni A, Blatt V, Pession A, Tallini G, Bertorelle R, Bartolini S, Calbucci F, Andreoli A, Frezza G, Leonardi M, Spagnolli F, Ermani M. MGMT promoter methylation status can predict the incidence and outcome of pseudoprogression after concomitant radiochemotherapy in newly diagnosed glioblastoma patients. J Clin Oncol. 2008 May 1;26(13):2192-7. doi: 10.1200/JCO.2007.14.8163. PMID 18445844